CLINICAL TRIAL: NCT05539872
Title: Comparison of the Pharmacokinetics (PK) and Pharmacodynamics (PD) Biosimilarity of Proposed Biosimilar Rapid-Acting Insulin Aspart (I004) and NovoLog After Single-Dose Subcutaneous Administration to Healthy Volunteers: A Single-Center Randomized, Double-blinded, Two-Treatment, Two-period, Two-sequence Crossover, Hyperinsulinemia-Euglycemic Clamp
Brief Title: Comparison of the Pharmacokinetics (PK) and Pharmacodynamics (PD) Biosimilarity of Proposed Biosimilar Rapid-Acting Insulin Aspart (I004) and NovoLog After Single-Dose Subcutaneous Administration to Healthy Volunteers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-I004-CL-B
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pharmacokinetics; Pharmacodynamics
Keywords: insulin aspart
MeSH Terms: interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin Aspart, I004 (Experimental): Participants who were dosed with I004
  Interventions: Drug: I004
- NovoLog (Active Comparator): Participants who were dosed with NovoLog
  Interventions: Drug: NovoLog

INTERVENTIONS:
Drug: I004 — Drug will be administered via subcutaneous injection into the abdominal wall of the peri-umbilical area with a dose of 0.2 units/kg based on the body weight measured at Treatment Period 1 under fasting condition.
  Other Names: Insulin Aspart, a rapid-acting human insulin analogue
  Arms: Insulin Aspart, I004
Drug: NovoLog — Drug will be administered via subcutaneous injection into the abdominal wall of the peri-umbilical area with a dose of 0.2 units/kg based on the body weight measured at Treatment Period 1 under fasting condition.
  Other Names: Insulin Aspart, a rapid-acting human insulin analogue
  Arms: NovoLog

SUMMARY:
This study is a randomized, double-blinded, two-treatment, two-period, two-sequence crossover pivotal Biosimilar study. The purpose of this study is to establish pharmacokinetic (PK) and pharmacodynamics (PD) biosimilarity of proposed biosimilar I004 and the US-approved NovoLog.

ELIGIBILITY:
Inclusion Criteria:

* Upon review, agree to participate and sign informed consent.
* Healthy male and female subjects ≥ 18 to ≤ 65 years of age.
* Body mass index (BMI) ≥ 18.5 to ≤ 29.9 kg/m2
* Weight ≥ 50 kg.
* Fasting plasma glucose of < 100 mg/dL (5.5 mmol/L) measured with YSI at site; one repeat test is allowed.
* HbA1c < 5.7%.
* Non-smoker for ≥ 3 months prior to Screening.
* Female candidates must be > 1 year post-menopausal, surgically sterile, or practicing a clinically acceptable form of birth control and confirmed by negative serum pregnancy test at Screening.

Exclusion Criteria:

* History of diabetes mellitus.
* Resting blood pressure (BP) > 140/90 mmHg or < 90/60 mmHg. Subjects BP may be re-checked.
* Participation in an investigational drug/device study within 30 days or 5 half-lives within the last dose of any study drug, whichever is longer.
* History of any serious adverse reaction or hypersensitivity to any of the investigational product components.
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders or abnormalities, or other major systemic disease that, according to the investigator, would unduly risk the subject's safety or may impact the conduct of the study.
* Subject shows evidence of significant active neuropsychiatric disease, including taking prescription medication for such diseases (including anti-depressant/anti-anxiety medication).
* Presence of clinically significant physical, laboratory, or ECG findings at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results, or may present a safety issue to that particular subject (laboratory results may be re-checked once on a separate day per Investigator discretion).
* Long QT syndrome or family history of long QT syndrome or corrected QT interval (QTcF) > 450 ms in men, > 470 ms in women at Screening.
* Liver function test results of AST and/or ALT ≥ 2.5 upper normal limit (ULN)
* Subject has a history of syncope.
* History of any major surgery within 6 months.
* History of any active infection, other than mild viral illness within 30 days prior to dosing.
* History of blood clots (e.g., deep vein thrombosis or embolism) or a frequent appearance in 1st degree relatives as judged by the Investigator.
* Known history or positive test of hepatitis B surface antigen (HBsAG), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibody.
* History of alcohol abuse as judged by the Investigator within approximately 1 year. Average weekly alcohol intake > 21 units/week (males) and > 14 units/week (females) or are unwilling to stop alcohol consumption from 24 hours prior to each dosing until discharged from the clinical research unit (CRU). Positive alcohol test at Screening. (One unit of alcohol equals about 250 mL of beer or lager, one glass of wine, or 20 mL of spirits).
* History of illicit drug abuse, including marijuana, within approximately 1 year or evidence of current use as judged by the Investigator. Positive drug test at Screening.
* Donation or loss of > 500 mL of blood within 56 days.
* Chronic use of over-the-counter or prescription medication within 7 or 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, or birth control methods [Desogestrel is not allowed]).
* Unable to comply with the safety monitoring requirements of this clinical study or is considered by the investigator to be an unsuitable candidate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Maximum Serum Insulin Aspart Concentration, CIAmax | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart
Area Under the Curve (AUC) of Insulin Aspart Serum Concentration from time 0 to 12 hours post-dose, AUCIA(0-12h) | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart. AUCIA(0-12h) will be calculated from the concentration curves.
Maximum Serum Human Insulin Concentration, CHImax | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Human Insulin
Area Under the Curve (AUC) of Human Insulin Serum Concentration from time 0 to 12 hours post-dose, AUCHI(0-12h) | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Human Insulin. AUCHI(0-12h) will be calculated from the concentration curves.
Maximum Glucose Infusion Rate, Gmax | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Area Under the Curve (AUC) for Glucose Infusion Rate from time 0 to 12 hours post-dose, AUCG(0-12h) | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response. AUCG(0-12h) will be calculated from the glucose infusion rate curves.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of Insulin Aspart Serum Concentration from time 0 to infinity, AUCIA(0-∞) | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart. AUCIA(0-∞) will be calculated from the concentration curves.
Area Under the Curve (AUC) of Insulin Aspart Serum Concentration from time 0 to 2 hours post-dose, AUCIA(0-2h) | From 60 minutes before dose until 2 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart. AUCIA(0-2h) will be calculated from the concentration curves.
Time of Maximum Insulin Aspart Serum Concentration, tIAmax | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart.
Apparent Clearance of Insulin Aspart, CL/F | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart.
Apparent Volume of Distribution of Insulin Aspart, Vz/F | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart.
Half-life of Insulin Aspart, t1/2 | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Insulin Aspart.
Time of Maximum Human Insulin Serum Concentration, tHImax | From 60 minutes before dose until 12 hours after dose
  Pharmacokinetic (PK) blood samples will be collected starting 60 minutes before dose and until 12 hours after dose. Serum will be isolated for analyzing the concentrations of Human Insulin.
Area Under the Curve (AUC) for Glucose Infusion Rate due to Insulin Aspart from time 0 to 12 hours post-dose, AUCGA(0-12h) | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response. AUCGA(0-12h) will be calculated from the glucose infusion rate curves.
Maximum Glucose Infusion Rate due to Insulin Aspart, GAmax | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Area Under the Curve (AUC) for Glucose Infusion Rate (GIR) from time 0 to the Time of Last Measureable GIR, AUCG(0-last) | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response. AUCG(0-last) will be calculated from the glucose infusion rate curves.
Area Under the Curve (AUC) for Glucose Infusion Rate from time 0 to 2 hours post-dose, AUCG(0-2h) | From drug administration until 2 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response. AUCG(0-2h) will be calculated from the glucose infusion rate curves.
Last Measureable Glucose Infusion Rate, Glast | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Time of Maximum Glucose Infusion Rate, tGmax | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Time of Glucose Infusion Start, tGonset | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Time of Last Measureable Glucose Infusion Rate, tGlast | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Time to Half of Maximum Glucose Infusion Rate (Gmax) Before Gmax Is Reached, tG50%early | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.
Time to Half of Maximum Glucose Infusion Rate (Gmax) After Gmax Is Reached, tG50%late | From drug administration until 12 hours after dose
  Participants will undergo a euglycemic clamp, where blood glucose concentration will be held at a constant target level by adjusting exogenous glucose infusion rate (GIR) following drug administration. GIR will be recorded for the duration of the euglycemic clamp and used to evaluate the Pharmacodynamic (PD) response.

CONTACTS AND LOCATIONS:
Locations (1):
- Amphastar Study Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Access to patient level data and supporting clinical documents may be requested by qualified researchers. Requests will be reviewed on the basis of scientific merit. Patient data will be de-identified to protect the privacy of trial patients in line with applicable laws and regulations.